CLINICAL TRIAL: NCT04190693
Title: IMCY-T1D-002: Long-term Follow-up Study of T1D Patients Previously Treated With IMCY-0098 or Placebo
Acronym: IMCY-T1D-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2018-003728-35
Record Dates: First submitted 2019-07-22; First posted 2019-12-09 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Long-term follow-up (LTFU), no study treatment administered.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment or Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follow-up (Placebo Comparator): No Investigational Medicinal Product (IMP) will be administered during this LTFU study. Patients received treatment with IMCY-0098 in the primary study (IMCY-T1D-001).
  Interventions: Drug: IMCY-0098 or placebo
- IMCY_0098 (Experimental): No Investigational Medicinal Product (IMP) will be administered during this LTFU study. Patients received treatment with IMCY-0098 in the primary study (IMCY-T1D-001).
  Interventions: Drug: IMCY-0098 or placebo

INTERVENTIONS:
Drug: IMCY-0098 or placebo — Long-term follow-up

SUMMARY:
This study is the follow-up of study IMCY-T1D 001 (EudraCT: 2016-003514-27, NCT03272269) in which patients with recent onset T1D have been treated with IMCY-0098 or placebo.

At the end of the primary 6 month study, patients will be proposed to enter this follow-up study to evaluate up to 12 months (V3 - Week 48) the safety, the immune responses and the clinical parameters.

The study involves a follow-up of 6 months after the end of the initial participation to the IMCY-T1D-001 study. Subjects will undergo visits at 24 weeks, 36 weeks and 48 weeks post first study product administration in study IMCY-T1D-001.

For each patient, the study comprises a total of 3 visits occurring over a period of approximately 24 weeks (from study entry). The patients will undergo planned assessments and procedures as outlined in the table of study procedures.

DETAILED DESCRIPTION:
In this Long-Term Follow-Up (LTFU) study, the below objectives will be assessed 36 and 48 weeks after the first injection of IMCY-0098 in the study IMCY-T1D-001, in patients treated with IMCY-0098 at three doses or placebo:

Primary Objective The primary objective of this study is to assess the long-term safety. Secondary Objective The secondary objective of this study is to evaluate the clinical response to IMCY-0098 by assessing disease activity.

Exploratory Objectives

* To evaluate the proinsulin-specific cytolytic CD4+ T cells induced by IMCY-0098
* To evaluate the impact of IMCY-0098 on autoreactive T-cell responses specific for autoantigens expressed by islet β-cells (proinsulin, GAD65, IGRP) on the longer-term.
* To evaluate the impact of IMCY-0098 on autoantibodies against GAD65, IA 2, ZnT8 and insulin
* Transcriptomic analysis on mRNA extracted from samples collected for Immunogenicity

ELIGIBILITY:
Inclusion Criteria:

* All patients who were treated with IMCY-0098 or placebo in the IMCY-T1D-001 clinical trial who are willing to participate to this long-term follow-up study.

Exclusion criteria:

* Ongoing pregnancy or lactation
* History of or current malignancy (except excised basal cell skin cancer)
* Primary or secondary immune deficiency disorders
* Human Immunodeficiency virus (HIV) infection.
* Ongoing treatment with immunosuppressive agents with the exception of topical or intra nasal corticosteroids.
* Treatment with an investigational drug within the past 3 months

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Van Rampelbergh, PhD, Study Director — Imcyse SA
Locations (19):
- Belgium (3):
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
- Hôpital Cochin, Paris, France
- Germany (2):
  - GWT-TUD GmbH, Dresden
  - Helmholtz Zentrum München - Deutsches Forschungszentrum für Gesundheit und Umwelt (GmbH), München
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - University Hospital Santaros Klinikos, Vilnius
- Sweden (2):
  - Clinical Trial Center, CTC, Gothenburg
  - ProbarE Stockholm, Stockholm
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff University, Cardiff
  - Royal Devon and Exeter NHS Trust, Exeter
  - Guy's and St. Thomas NHS Trust, London
  - St. Bartholomew's Hospital (Barts Health NHS Trust), London
  - Newcastle University, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Rampelbergh J, Achenbach P, Leslie RD, Ali MA, Dayan C, Keymeulen B, Owen KR, Kindermans M, Parmentier F, Carlier V, Ahangarani RR, Gebruers E, Bovy N, Vanderelst L, Van Mechelen M, Vandepapeliere P, Boitard C. First-in-human, double-blind, randomized phase 1b study of peptide immunotherapy IMCY-0098 in new-onset type 1 diabetes. BMC Med. 2023 May 24;21(1):190. doi: 10.1186/s12916-023-02900-z. PMID 37226224

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patients having received 50 μg IMP (2x subcutaneous [s.c.] injections of 25 μg [100 μL each]) + 3x 25 μg IMP (each as 2x s.c. injections of 12.5 μg [50 μL each]) in study 2016-003514-27
- Cohort 2: Patients having received 150 μg IMP (2x s.c. injections of 75 μg [300 μL each]) + 3x 75 μg IMP (each as 2x s.c injections of 12.5 μg [150 μL each]) in study 2016-003514-27
- Cohort 3: Patients having received 450 μg IMP (2x s.c. injections of 225 μg [900 μL each]) + 3x 225 μg IMP (each as 2x s.c injections of 112.5 μg [450 μL each]) in study 2016-003514-27
- Placebo: Patients having received Placebo in study 2016-003514-27
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Started | 4 | 7 | 12 | 7
Completed | 4 | 7 | 12 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo | Total
Number analyzed (Participants) | 4 | 7 | 12 | 7 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 12 | 7 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (2.7) | 26.1 (4.3) | 25.1 (4.8) | 26.0 (3.9) | 25.5 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender categorical: Female | 1 | 2 | 3 | 3 | 9
  Gender categorical: Male | 3 | 5 | 9 | 4 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Time Frame: Throughout the study period (24weeks)
Measure: Number; unit: Number of AE
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 4 | 7 | 12 | 7
Number of AE | 5 | 6 | 10 | 4

2. Primary Outcome: Serious Adverse Events
Time Frame: Throughout the study period (24 weeks)
Measure: Number; unit: Number of SAE
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 4 | 7 | 12 | 7
Number of SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period (24 weeks)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 2/4 | 3/7 | 6/12 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=7) | Cohort 3 (N=12) | Placebo (N=7)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adbominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal ski infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT04190693/Prot_SAP_000.pdf